CLINICAL TRIAL: NCT02450019
Title: Protective Ventilation in Neurosurgery, a Pilot Study
Acronym: NeuroVentOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Marco Gemma, MD Anaesthesist, IRCCS San Raffaele
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 22/INT/2015
Record Dates: First submitted 2015-05-09; First posted 2015-05-21 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Nervous System Neoplasms
MeSH Terms: conditions — Nervous System Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Traditional to protective ventilation (Other): Traditional ventilation will be set with 9 ml/kg with predicted body weight of tidal volumes and no PEEP. Arterial CO2 partial pressure will be maintained between 30 and 35 mmHg. After intracranial pressure measurement ventilation will be switched to protective.
  Interventions: Procedure: Traditional to protective ventilation
- Protective to traditional ventilation (Other): Protective ventilation will be set with 7 ml/kg tidal volume, 5 cm H2O PEEP, and 0.4 inspired O2 fraction (FiO2). Arterial CO2 partial pressure will be maintained between 30 and 35 mmHg. After intracranial pressure measurement ventilation will be switched to traditional.
  Interventions: Procedure: Protective to traditional ventilation

INTERVENTIONS:
Procedure: Traditional to protective ventilation — Traditional ventilation will be set with 9 ml/kg with predicted body weight of tidal volumes and no PEEP and switched to protective ventilation after intracranial pressure measurement.
  Other Names: Traditional to protective
  Arms: Traditional to protective ventilation
Procedure: Protective to traditional ventilation — Protective ventilation will be set with 7 ml/kg tidal volume, 5 cm H2O PEEP, and 0.4 inspired O2 fraction (FiO2), and switched to traditional ventilation after intracranial pressure measurement.
  Arms: Protective to traditional ventilation

SUMMARY:
The purpose of this study is to assess the effect size and variability of dural tension measured as intracranial pressure (ICP) below the dura of the surgical field in patients undergoing elective supra-tentorial surgery for brain neoplasms in patients alternatively ventilated with traditional high-volume-no-PEEP ventilation and protective low-volume-low-PEEP ventilation.

DETAILED DESCRIPTION:
The role of mechanical ventilation in patients undergoing general anesthesia is worldwide well known but it has been associated with dangerous effects such as pulmonary complications, increasing postoperative morbidity and mortality. Lung-protective ventilation using low tidal volume and positive end-expiratory pressure (PEEP), can reduce morbidity and mortality in patients with acute respiratory distress syndrome and is now considered a strong recommendation in patients undergoing general anesthesia. At the moment there are no guidelines that define which kind of ventilation should be used.

Patients without acute lung injury are still ventilated with large -and perhaps too large- tidal volumes. A recent multicenter randomized controlled trial has concluded that the use of a lung-protective ventilation strategy in intermediate-risk and high-risk patients undergoing major abdominal surgery was associated with improved clinical outcomes and reduced health care utilization . A multicentre randomized controlled trial on mechanical ventilation during general anesthesia for open abdominal surgery has concluded that an intraoperative protective ventilation strategy should include a low tidal volume and low PEEP, without recruitment maneuvers. In 52 patients undergoing general anesthesia for open thoracic surgery lung protective ventilation was associated with better intraoperative and postoperative oxygenation, and shorter duration of postoperative mechanical ventilation from ICU admission to its withdrawal.

In conclusion protective ventilation, with low tidal volumes and low PEEP, seems to be the gold standard for intra-operative mechanical ventilation during general anesthesia.

Mechanical ventilation represents an important tool to obtain cerebral de-bulking during neurosurgery by maintaining moderate hypocapnia and positive intra-thoracic pressure the lowest possible. For these reasons the application of PEEP with high tidal volume has been historically seen as unfavourable by neuro-anesthesiologists and neurosurgeons fearing transmission to intracranial compartment of high venous pressure values with consequent brain swelling and eventually cerebral perfusion pressure reduction.

Nevertheless, recent studies suggested that in patients with traumatic brain injury (TBI) PEEP seems to be well tolerated without deleterious intracranial effect and its role in the context of a protective ventilation protocol associated with low tidal volume, so with low expected intra-thoracic pressures, has never been studied in patients undergoing to general anesthesia for intracranial surgery of neoplasms.

The traditional high-volume-no-PEEP ventilation strategy, called this way because it consists of an higher tidal volumes than protective ventilation and no PEEP, in neurosurgery should be compared with the recently proposed protective ventilation in order to eventually assess possible differences on respiratory and neurological outcomes. At this purpose a pilot study is needed to determine the effect size and variability of possible differences in dural tension between the two ventilation strategies.

Null hypothesis: Shifting from traditional ventilation protocol to a protective one during general anesthesia does not change levels of dural tension in patients undergone to elective neurosurgery for brain neoplasms.

To determine the effect size and variability of dural tension differences in patients undergoing intracranial neurosurgery and ventilated with either traditional or protective ventilation.

Mono-centric, double blind, 1:1 randomized, 2x2 crossover clinical trial. Patients will be randomized to receive either traditional or protective ventilation as the first ventilation. Randomization will be performed by a computer generated sequence. The results of the randomization will be transferred in sealed envelopes, one for each patient. When the patient will be randomized in the study, the envelop will be open and the piece of information about the randomization present in the envelop will be followed by the operating room anesthesiologist.

ELIGIBILITY:
Inclusion Criteria:

Elective surgical removal of a supra-tentorial neoplasm conditioning mass effect defined as:

* Median line shift at preoperative CT scan ≥ 5mm
* Cortical brain effacement at preoperative CT scan

Exclusion Criteria:

* Age < 18 yrs or > 80 yrs.
* BMI > 30
* Pregnancy.
* Refusal to sign the informed consent.
* Emergency surgery.
* Respiratory co-morbidities (clinical evidence or history of COPD, asthma, interstitial pneumopathies, previous thoracic surgery).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-05; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Intracranial pressure measured in mmHg | Outcome 1 is assessed before the incision of dura mater (mean 1 hour).
  Primary endpoint: to assess the effect size and variability of dural tension measured as intracranial pressure (ICP) below the dura of the surgical field in patients undergoing elective supra-tentorial surgery for brain neoplasms in patients alternatively ventilated with traditional high-volume-no-PEEP ventilation and protective low-volume-low-PEEP ventilation.

SECONDARY OUTCOMES:
Dural tension measured by a two point scale (acceptable/unacceptable). | Outcome 2 is assessed before the incision of dura mater (mean 1 hour).
  Secondary endpoints: subjective assessment of dural tension by the attending neurosurgeon quantified as "acceptable tension" or "unacceptable tension" at the end of crossover.

CONTACTS AND LOCATIONS:
Locations (1):
- S. Raffaele Hospital, Milan, MI, Italy